CLINICAL TRIAL: NCT07164612
Title: The Effectiveness of Occupation-based Bilateral Arm Training on Motor Functions and Activity Participation Among Stroke Survivors During Inpatient Rehabilitation. A Randomized Control Trial
Brief Title: The Effectiveness of Occupation-based Bilateral Arm Training on Motor Functions and Activity Participation Among Stroke Survivors During Inpatient Rehabilitation.
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hamad Medical Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MRC-01-25-298
Record Dates: First submitted 2025-09-02; First posted 2025-09-10 (Actual); Last update posted 2025-09-22 (Actual); Status verified 2025-09

CONDITIONS: Stroke
Keywords: Stroke; Occupations; Occupation-based intervention; Occupational Therapy; Motor Activity; Motor Skills; Patient Participation
MeSH Terms: conditions — Stroke; Motor Activity; Patient Participation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Data Analyst
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- OBBT group (Experimental): Participants in the experimental group will receive face- to- face individual 30 minutes OBBT program in addition to conventional therapy. These 30 -minute OBBT session will be added to the standard conventional therapy sessions (90 minutes).
  Interventions: Other: Occupation-Based Bilateral Upper Limb Training (OBBT)
- Conventional Therapy (control group) (Other): Participants in the control group will receive conventional therapy consisting of standard rehabilitation approaches for upper limb impairments.
  Interventions: Other: Conventional therapy group

INTERVENTIONS:
Other: Occupation-Based Bilateral Upper Limb Training (OBBT) — Intervention sessions for experimental group will be conducted 5 times per week over 6 weeks. OBBT will be used to engage both upper limbs simultaneously in simulate real-life functional tasks which tailored to individual needs, focusing on improving the patient's ability to perform daily activities such as dressing, washing, and cooking. The training will emphasize occupation-specific repetitive practice for at least two selected occupations and encouraged active participation of both hands during functional tasks to improve use of both upper limb motor functions and activity participation. Additionally, it will seek to support stroke survivors in their pursuit of an independent, productive, and functional recover.
  Arms: OBBT group
Other: Conventional therapy group — Conventional therapy includes passive and active range of motion exercises, strengthening exercises, basic functional activities and mobility training, and activities designed to improve muscle tone and mobility in the affected upper limb among stroke survivors. The conventional therapy sessions will be delivered 5 times per week for 90 minutes over 6 weeks. Therapy sessions will be individualized to the participant's needs and will be provided by senior occupational therapists.
  Arms: Conventional Therapy (control group)

SUMMARY:
People with stroke often experience limitations in motor functions and activity participation. Occupation-based bilateral upper limb training (OBBT) using occupations as meaningful daily activities, and as part of the therapy. The activities in OBBT are tailored to the patient's life with the goal of boosting motivation and engagement to enhance activity performance and participation. This study is a randomized control trial that aims to explore the effect of OBBT along with the conventional therapy in comparison with the conventional therapy alone on motor functions and activity participation among stroke survivors in inpatient rehabilitation setting. This study will be conducted in Qatar Rehabilitation Institute, Hamad Medical Corporation, Doha, Qatar. Participants will be allocated randomly to either the OBBT group or the conventional therapy group. Participants in the OBBT group will receive 30 minutes OBBT program in addition to conventional therapy (90 minutes). Intervention sessions will be conducted 5 times per week over 6 weeks. The participants in the conventional therapy group will receive only the conventional therapy (90 minute). All participants will be assessed using the outcome measure immediately the day after completing the last intervention session at 4th week and 6th week.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosed with first ischemic or hemorrhagic stroke by medical physician
2. Stroke onset ≤ 6 months
3. Both males and females with age 18-65 years
4. Cognitive functions within normal and mild deficit (MMSE ≥ 22)
5. With arm and hand upper extremity Brunnstrom stage of >3
6. Free of any other neurological diseases.

Exclusion Criteria:

1. participants with previous stroke
2. musculoskeletal disease or sever pain affecting the upper extremities
3. participant who have taken part in another rehabilitative research
4. sever visual neglect or visual field deficit.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2025-09 (Estimated); Primary Completion 2027-04 (Estimated); Study Completion 2027-09 (Estimated)

PRIMARY OUTCOMES:
Fugl-Meyer Assessment (FMA) | At baseline, immediately post 4th weeks, and 6th week of the intervention.
  More than 80% of studies use the Fugl-Meyer Assessment, making it the most popular outcome measure for evaluating upper limb motor function recovery after stroke. The assessment consists18 items for the shoulder, elbow, 5 items for the wrist, 7 items for the hand and fingers, and 3 items for upper extremity coordination. The total Fugl-Meyer Assessment (FMA) motor function score for the upper extremity is 66, with higher scores indicating greater motor performance.

SECONDARY OUTCOMES:
Action Research Arm Test (ARAT) | It will be conducted at baseline, immediately post 4th weeks, and 6th week of the intervention.
  To examine the motor function for the paretic side. Action Research Arm Test consists 19 items distributed into 4 subscales of grasp, grip, pinch and gross movement. The total score on the Action Research Arm Test (ARAT) is 57, with higher scores indicating better motor performance.
Functional independence measure (FIM) | At baseline, immediately post 4th weeks, and 6th week of the intervention.
  Functional Independent Measure (FIM) will be used to evaluate functional independence in activities such as self-care, sphincter control, transfer, locomotion, communication, and social cognition. It includes 18 items total, with a maximum score of 7 and a minimum score of 1, for a total score of 126. Higher score means more independent.
Stroke Impact Scale (SIS) | At baseline, immediately post 4th weeks, and 6th week of the intervention.
  Stroke Impact Scale (SIS) will be used to detect the progress in stroke recovery. It includes 64 items into 8 parts including, strength, Activities of Daily Living, Instrumental Activities of Daily Living, mobility, hand function, memory and communication, emotion and participant. The Stroke Impact Scale (SIS) is a continuous measure ranging from 0 to 100, where 0 indicates no recovery and 100 indicates full recovery. Higher scores reflect greater perceived recovery.
Canadian Occupational Performance Measure (COPM) | At baseline, immediately post 4th weeks, and 6th week of the intervention.
  Canadian Occupational Performance Measure (COPM) will be used to measure occupational performance ability. It includes a four stage, semi-constructive meeting session, participants will be asked to consider their goals, needs, and expectations for their daily lives. Performance and satisfaction with the chosen activity will then be measured on a 10 point scale with higher score means a greater performance and satisfaction.
  In this study participant's choice of occupation-based activities and improvement in their performance and satisfaction, before and after the intervention, will be assessed using COPM.

CONTACTS AND LOCATIONS:
Locations (1):
- Hamad Medical Corporation\ Qatar Rehabilitation Institute, Doha, Qatar

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Dembele J, Triccas LT, Amanzonwe LER, Kossi O, Spooren A. Bilateral versus unilateral upper limb training in (sub)acute stroke: A systematic and meta-analysis. S Afr J Physiother. 2024 Jan 23;80(1):1985. doi: 10.4102/sajp.v80i1.1985. eCollection 2024. PMID 38322652
- [Background] Kim SH, Park JH. The Effect of Occupation-Based Bilateral Upper Extremity Training in a Medical Setting for Stroke Patients: A Single-Blinded, Pilot Randomized Controlled Trial. J Stroke Cerebrovasc Dis. 2019 Dec;28(12):104335. doi: 10.1016/j.jstrokecerebrovasdis.2019.104335. Epub 2019 Sep 30. PMID 31582271
- [Background] Meng G, Meng X, Tan Y, Yu J, Jin A, Zhao Y, Liu X. Short-term Efficacy of Hand-Arm Bimanual Intensive Training on Upper Arm Function in Acute Stroke Patients: A Randomized Controlled Trial. Front Neurol. 2018 Jan 19;8:726. doi: 10.3389/fneur.2017.00726. eCollection 2017. PMID 29403422
- [Background] Renner CIE, Brendel C, Hummelsheim H. Bilateral Arm Training vs Unilateral Arm Training for Severely Affected Patients With Stroke: Exploratory Single-Blinded Randomized Controlled Trial. Arch Phys Med Rehabil. 2020 Jul;101(7):1120-1130. doi: 10.1016/j.apmr.2020.02.007. Epub 2020 Mar 4. PMID 32145277
- [Background] Stoykov ME, Lewis GN, Corcos DM. Comparison of bilateral and unilateral training for upper extremity hemiparesis in stroke. Neurorehabil Neural Repair. 2009 Nov;23(9):945-53. doi: 10.1177/1545968309338190. Epub 2009 Jun 16. PMID 19531608
- [Background] Summers JJ, Kagerer FA, Garry MI, Hiraga CY, Loftus A, Cauraugh JH. Bilateral and unilateral movement training on upper limb function in chronic stroke patients: A TMS study. J Neurol Sci. 2007 Jan 15;252(1):76-82. doi: 10.1016/j.jns.2006.10.011. Epub 2006 Nov 28. PMID 17134723